CLINICAL TRIAL: NCT01309165
Title: Exploring the Efficacy of Combined Task-Specific and Cognitive Strategy Training in Subacute Stroke: A Phase II Clinical Trial.
Brief Title: Exploring the Efficacy of Combined Task-Specific and Cognitive Strategy Training in Subacute Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. John's Rehab Hospital (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other); Washington University School of Medicine (Other); University of Toronto (Other)
Responsible Party: Principal Investigator, Sara McEwen, Research Scientist, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIHR 230433
Record Dates: First submitted 2011-03-04; First posted 2011-03-07 (Estimated); Results first posted 2019-02-08 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2018-09

CONDITIONS: Stroke
Keywords: stroke; cognition; cognitive strategies; motor skill acquisition; participation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CO-OP (Experimental): CO-OP, a client-centred, performance-based, problem solving approach has 7 key features including: client-chosen goals, dynamic performance analysis, cognitive strategy use, guided discovery, and a specific 10 one-hour sessions intervention format. Participants randomized to the CO-OP group will continue to receive usual out-patient services, such as physiotherapy or speech-language therapy, but will receive CO-OP instead of usual occupational therapy.
  Interventions: Behavioral: CO-OP
- Standard Occupational Therapy (Active Comparator): Participants randomized to the SOT group will receive usual out-patient rehabilitation services, with slight modifications. Specifically, a research assistant will administer the COPM to assist participants to self-select 4 personally meaningful skills. The treating SOT occupational therapists will be asked to log the activities completed in each session, and the amount of time spent in therapy.
  Interventions: Behavioral: Standard Occupational Therapy

INTERVENTIONS:
Behavioral: CO-OP — CO-OP, a client-centred, performance-based, problem solving approach has 7 key features including: client-chosen goals, dynamic performance analysis, cognitive strategy use, guided discovery, and a specific 10-session intervention format. The client and the therapist work together, using the Canadian Occupational Performance Measure (COPM), to select 3 skills and establish baseline skill performance. In the second meeting, when CO-OP actually begins, the approach is introduced to the client and the global cognitive strategy (GOAL-PLAN-DO-CHECK) is learned. In all subsequent sessions this strategy is used as the main problem-solving framework to facilitate skill acquisition.
  Arms: CO-OP
Behavioral: Standard Occupational Therapy — Participants randomized to the SOT group will receive usual out-patient rehabilitation services, with slight modifications. Specifically, a research assistant will administer the COPM to assist participants to self-select 4 personally meaningful skills. The treating SOT occupational therapists will be asked to log the activities completed in each session, and the amount of time spent in therapy.
  Arms: Standard Occupational Therapy

SUMMARY:
Novel stroke rehabilitation approaches, such as task-specific training (TST), have shown promise in improving stroke recovery components such as basic mobility and activities of daily living; however, evidence suggests these improvements are not generalized and transferred to home, community, or work settings, and usually do not impact overall participation outcomes. Further, these treatments are very intense, with total treatment times as high as 30 to 60 hours, making them clinically or economically unfeasible in many settings. In contrast, approaches incorporating cognitive strategy training have shown great promise to not only improve functional activity performance in people living with stroke, but also to facilitate generalization and transfer beyond the clinical setting, and to do so in 10 to 15 treatment hours. Cognitive Orientation to daily Occupational Performance (CO-OP) is an established treatment approach that uses cognitive strategies in combination with TST. Evidence from other research groups and findings from our own participant interview data indicate that the approach may be even more effective if introduced much earlier in the rehabilitation process, however, CO-OP has not yet been tested in this sub-acute population. Therefore, the specific project goals are: 1. To refine the CO-OP treatment approach for use with people less than three months post stroke; 2. To evaluate, in a Phase II clinical trial, the preliminary efficacy of the refined protocol compared to standard occupational therapy on immediate and longer-term skill performance and participation; 3. To determine effect sizes for power calculations for a future Phase III clinical trial to test the new protocol versus contemporary treatment. The research approach consists of Part 1, Protocol Refinement, and Part 2, Exploratory Phase II Clinical Trial.

DETAILED DESCRIPTION:
Activity and participation limitations occur in the majority of those living with the effects of stroke. Novel stroke rehabilitation approaches, such as task-specific training (TST), have shown promise in improving recovery components such as basic mobility and activities of daily living; however, evidence suggests these improvements are not generalized and transferred to home, community, or work settings, and usually do not impact overall participation outcomes. Further, these treatments are very intense, with total treatment times as high as 30 to 60 hours, making them clinically or economically unfeasible in many settings. In contrast, approaches incorporating cognitive strategy training have shown great promise to not only improve functional activity performance in people living with stroke, but also to facilitate generalization and transfer beyond the clinical setting, and to do so in 10 to15 treatment hours.

Cognitive Orientation to daily Occupational Performance (CO-OP) is an established treatment approach that uses cognitive strategies in combination with TST. Cognitive strategies are learning strategies that are goal directed and derived from cognitive executive functions such as initiation, planning, and error detection, that support early and mid phase skill acquisition. TST is based on the principles of motor learning, such as optimal provision of feedback and practice schedules, and involves repetitive practice of specific tasks, skills, or activities. Research from the investigators lab demonstrated that CO-OP is associated with functional skill acquisition, retention, and generalization and transfer of skills beyond the rehabilitation setting in adults more than one year post-stroke. Evidence from other research groups and findings from our own participant interview data indicate that the approach may be even more effective if introduced much earlier in the rehabilitation process, however, CO-OP has not yet been tested in this sub-acute population. Therefore, the specific project goals are:

1. To refine the CO-OP treatment approach for use with people less than three months post stroke;
2. To evaluate, in a Phase II clinical trial, the preliminary efficacy of the refined protocol compared to TST alone on immediate and longer-term skill performance and participation;
3. To determine effect sizes for power calculations for a future Phase III clinical trial to test the new protocol vs. contemporary treatment.

The research approach consists of Part 1, Protocol Refinement, and Part 2, Exploratory Phase II Clinical Trial. Part 1 addresses the first project goal of refining CO-OP for use with people less than three months post stroke. In Part 1, three to four adults, less than three months post stroke, will be recruited. The CO-OP protocol will be iteratively modified as necessary based on the experience with each participant, the treating therapists' logs, treatment outcome data, and research team consensus.

Part 2, Exploratory Phase II Clinical trial with Control Arm, will address the second and third project goals. Part 2 will make use of the treatment protocol refinements from Part 1. Based on data from our studies with more chronic patients, an estimated sample size of 28 patients, 14 per group, will provide 82% power to detect a treatment difference of 1.3 units on the Canadian Occupational Performance Measure (COPM), standard deviation 1.15. The main study outcomes will be changes in performance quality of both trained and untrained skills, as measured by the participant-rated COPM and the observer-rated Performance Quality Rating Scale (PQRS); and changes in participation, as measured by the Participation Domain of the Stroke Impact Scale (SIS). Data analysis will consist of descriptive statistics and between- and within-group differences. Variability in outcome measures will be coupled with estimates of clinically meaningful effect size to conduct sample size calculations for the future Phase III clinical trial. As well, data informative to feasibility will be examined, such as recruitment rate, attrition, mean number of sessions completed, and treatment satisfaction ratings.

The innovation of this proposal is that it will enhance stroke rehabilitation and important long-term functional and participation stroke outcomes through the efficient mechanism of adding cognitive strategy use to existing TST-based programs. The significance is high, in that those with stroke are at high risk for declining participation and increased resource utilization.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years of age or greater
* Admitted to out-patient rehabilitation post ischemic stroke

Exclusion Criteria:

* more than 6 months post stroke onset
* those not requiring occupational therapy
* hemorrhagic stroke
* neurological diagnoses other than stroke
* major psychiatric illness
* moderate or severe aphasia (NIH Stroke Scale aphasia rating of 2 or more)
* dementia (Mini Mental State Exam scores of 24 or less)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara E McEwen, PhD, Principal Investigator — University of Toronto
Locations (2):
- Rehabilitation Institute of St. Louis, St Louis, Missouri, United States
- St. John's Rehab; Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Result] McEwen S, Polatajko H, Baum C, Rios J, Cirone D, Doherty M, Wolf T. Combined Cognitive-Strategy and Task-Specific Training Improve Transfer to Untrained Activities in Subacute Stroke: An Exploratory Randomized Controlled Trial. Neurorehabil Neural Repair. 2015 Jul;29(6):526-36. doi: 10.1177/1545968314558602. Epub 2014 Nov 21. PMID 25416738
- [Result] Wolf TJ, Polatajko H, Baum C, Rios J, Cirone D, Doherty M, McEwen S. Combined Cognitive-Strategy and Task-Specific Training Affects Cognition and Upper-Extremity Function in Subacute Stroke: An Exploratory Randomized Controlled Trial. Am J Occup Ther. 2016 Mar-Apr;70(2):7002290010p1-7002290010p10. doi: 10.5014/ajot.2016.017293. PMID 26943113

RESULTS

PARTICIPANT FLOW:
Groups:
- CO-OP: CO-OP: CO-OP, a client-centred, performance-based, problem solving approach has 7 key features including: client-chosen goals, dynamic performance analysis, cognitive strategy use, guided discovery, and a specific 10-session intervention format. The client and the therapist work together, using the Canadian Occupational Performance Measure (COPM), to select 3 skills and establish baseline skill performance. In the second meeting, when CO-OP actually begins, the approach is introduced to the client and the global cognitive strategy (GOAL-PLAN-DO-CHECK) is learned. In all subsequent sessions this strategy is used as the main problem-solving framework to facilitate skill acquisition.Participants randomized to the CO-OP group will continue to receive usual out-patient services, such as physiotherapy or speech-language therapy, but will receive CO-OP instead of usual occupational therapy.
Period: Overall Study
Arm/Group | CO-OP | Standard Occupational Therapy
Started | 19 | 16
Received Allocated Intervention | 16 | 14
Included in Primary Analysis | 14 | 12
Completed | 13 | 9
Not Completed | 6 | 7
Not completed — Lost to Follow-up | 4 | 3
Not completed — Return to work | 1 | 2
Not completed — Left country | 0 | 1
Not completed — No transportation | 0 | 1
Not completed — Admitted to hospital for second stroke | 1 | 0

BASELINE CHARACTERISTICS:
Population: There were 35 participants enrolled in the study and baseline characteristics were collected for all. Of those, 30 received the allocated intervention (19 for CO-OP and 16 for Standard OT). Due to participant withdrawal, 26 were included in the primary analysis (14 for CO-OP and 12 for Standard OT).
Groups:
- Total: Total of all reporting groups
Arm/Group | CO-OP | Standard Occupational Therapy | Total
Number analyzed (Participants) | 19 | 16 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (14) | 54.4 (14) | 56.1 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 13 | 9 | 22
Region of Enrollment [Number; unit: participants]
  Canada | 8 | 7 | 15
  United States | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Performance Quality Rating Scale (PQRS)
Description: The Performance Quality Rating Scale (PQRS) rates performance on a 10-point scale, with a score of 1 indicating "can't do the skill at all" and 10 indicating "does the skill very well". Inter-rater reliability in the stroke population has been estimated at 0.71 (ICC). An independent observer rates performances from video recorded trials of each skill at all assessment points.
  Data reported are the average of participants' trained and untrained change scores e.g. Time 2 minus Time 1 and Time 3 minus Time 1.
  Therapist logs and institutional patient records were reviewed to establish which self-selected activities were trained during the occupational rehabilitation program. A self-selected activity was considered trained if there was any indication of practicing all or part of it or any and indication of discussions or education concerning the activity. If no evidence of training was found it was considered untrained.
Time Frame: A) Time 1- Baseline, B) Time 2- post-intervention (approx. 6 weeks from baseline), C) Time 3- 3 month follow-up (approx. 17 weeks from baseline)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CO-OP | Standard Occupational Therapy
Number analyzed (Participants) | 14 | 12
units on a scale
  Time 2 - 1 Mean Change - Trained | 2.9 (1.4) | 1.8 (2.9)
  Time 3 - 1 Mean Change - Trained | 4.5 (1.7) | 1.5 (2.2)
  Time 2 - 1 Mean Change - Untrained | 2.9 (1.4) | 0.5 (2.5)
  Time 3 - 1 Mean Change - Untrained | 3.6 (2.3) | 1.5 (2.0)

2. Secondary Outcome: Change From Baseline in Canadian Occupational Performance Measure (COPM)
Description: The Canadian Occupational Performance Measure (COPM) is a standardized instrument for eliciting performance issues from the client perspective, and for capturing perceived changes in performance over time.The COPM will be used to elicit participant-selected goals. It will also be used to rate self-perceived performance and performance satisfaction for each goal. Scores range from 1 to 10 (higher is better).
  Data reported are the average of participants' trained and untrained change scores e.g. Time 2 minus Time 1 and Time 3 minus Time 1.
  Therapist logs and institutional patient records were reviewed to establish which self-selected activities were trained during the occupational rehabilitation program. A self-selected activity was considered trained if there was any indication of practicing all or part of it or any and indication of discussions or education concerning the activity. If no evidence of training was found it was considered untrained.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CO-OP | Standard Occupational Therapy
Number analyzed (Participants) | 14 | 12
units on a scale
  Time 2-1 Mean Change Score - Performance - Trained | 1.5 (3) | 2.3 (2.1)
  Time 3-1 Mean Change Score - Performance - Trained | 2.9 (1.8) | 2.3 (2.5)
  Time 2-1 Mean Change Score - Performance-Untrained | 1.3 (3.1) | 1.9 (2.3)
  Time 3-1 Mean Change Score - Performance-Untrained | 3.1 (2.7) | 2.4 (2.5)
  Time 2-1 Mean Change Score - Satisfaction- Trained | 1.9 (2.8) | 1.8 (2.3)
  Time 3-1 Mean Change Score - Satisfaction- Trained | 3.2 (1.8) | 3.7 (3.3)
  Time 2-1 Mean Change Score- Satisfaction-Untrained | 1.5 (3.3) | 1.7 (2.1)
  Time 3-1 Mean Change Score- Satisfaction-Untrained | 3.2 (3) | 2.8 (2.3)

3. Secondary Outcome: Change From Baseline in Stroke Impact Scale (SIS) Participation Domain
Description: The Stroke Impact Scale (SIS) is a stroke-specific health status measure. The scale is comprised of nine domains, of which we are using one, the Participation Domain.
  Scores range from 0-100 (higher is better).
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CO-OP | Standard Occupational Therapy
Number analyzed (Participants) | 14 | 12
units on a scale
  Time 2 Mean Score | 47.9 (16.8) | 54.6 (13.7)
  Time 3 Mean Score | 56.6 (16.7) | 56.9 (13.3)
  Time 3-1 Mean Change Score | 8.0 (9.9) | 1.9 (12.5)

4. Secondary Outcome: Change From Baseline in Activity Card Sort (ACS)
Description: The Activity Card Sort (ACS) is a client-centred interview based instrument that identifies participation in instrumental, social, and high- and low- demand physical leisure activities. A sorting methodology is used to identify whether or not the person performed the activity before their stroke and the person identifies the activities that are most important to them. The properties of ACS have been tested in various populations and there is evidence for internal consistency, construct, concurrent, and discriminant validity.
  Data reported are the average of participants' trained and untrained change scores e.g. Time 2 minus Time 1 and Time 3 minus Time 1.
Time Frame: A) Time 2- post-intervention (approx. 6 weeks from baseline), B) Time 3- 3 month follow-up (approx. 17 weeks from baseline)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CO-OP | Standard Occupational Therapy
Number analyzed (Participants) | 14 | 12
units on a scale
  Time 2 Mean Total | 34.4 (12.7) | 28.1 (11.6)
  Time 3 Mean Total | 37.4 (13.0) | 29.6 (7.2)

ADVERSE EVENTS:
Arm/Group | CO-OP | Standard Occupational Therapy
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/16
Other Adverse Events (participants affected / at risk) | 0/19 | 0/16

LIMITATIONS AND CAVEATS:
Statistical analysis was limited to univariate procedures and could not control for the effect of confounders; the usual care control was unstandardized; the study included a short follow-up period of 3 months after the post-intervention session.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No